CLINICAL TRIAL: NCT06727929
Title: The Effect of Non-surgical Periodontal Treatment on Gingival Crevicular Fluid Dickkoff-1(Dkk-1) and Secreted Frizzled Related Protein 5 (sFRP5) Levels
Brief Title: The Effect of Non-surgical Periodontal Treatment on Dickkoff-1 and Secreted Frizzled Related Protein-5 Levels
Status: Active, not recruiting | Type: Observational
Sponsor: Cumhuriyet University (Other)
Collaborators: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Sukran Acipinar, Ass.Prof., Cumhuriyet University
Other Study IDs: SCU
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Periodontal Inflammation; Alveolar Bone Loss; Periodontal Diseases
Keywords: Dickkopf-1; secreted Frizzled Related Protein 5; Gingival crevicular fluid
MeSH Terms: conditions — Alveolar Bone Loss; Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Periodontally Healthy: PD ≤3 mm, fullmouth bleeding scores (BOP) % <10, no CAL and radiologic bone loss
  Interventions: Diagnostic Test: Collection of gingival crevicular fluid, ELISA
- Gingivitis: PD ≤3 mm, % BOP >30, no CAL(due to periodontal disease) and radiologic bone loss
  Interventions: Diagnostic Test: Collection of gingival crevicular fluid, ELISA
- Periodontitis: These individuals had a minimum of two non-adjacent teeth with sites with PD ≥6 mm, CAL ≥5 mm, BOP ≥30%, tooth loss due to periodontitis ≤4 teeth, the alveolar bone loss at radiographs extending to middle or apical third of the root, the presence of consistent amounts of plaque biofilm/calculus deposits commensurate with the severity of periodontal tissue breakdown, the proportion of percentage bone loss to age values were between 0.25 and 1
  Interventions: Diagnostic Test: Collection of gingival crevicular fluid, ELISA

INTERVENTIONS:
Diagnostic Test: Collection of gingival crevicular fluid, ELISA — GCF samples were collected at baseline and at the 6-8 -week follow-up appointment after non-surgical periodontal treatment . After removing the supragingival plaque from the interproximal surfaces with sterile curettes, these sample surfaces were isolated with cotton rolls and slightly air-dried to avoid contamination. Standardized paper strips were inserted 1 to 2 mm into the gingival sulcus and held for 30 seconds to collect GCF. Strips contaminated with blood or saliva were discarded and not evaluated. The paper strips were transferred to a precalibrated Periotron 8000 device to measure the fluid volume. Paper strips were placed in sterile Eppendorf tubes and stored at -80C, until laboratory analysis. The level of GCF Dkk-1 and sFRP5 levels was measured by ELISA using commercial kits.

SUMMARY:
Periodontitis is a condition that is defined by microbial-associated, host-induced inflammation, which ultimately results in the loss of periodontal attachment.Periodontal clinical parameters are the most reliable indicators of periodontal disease; however, they provide information about past tissue destruction and are insufficient for predicting future periodontal disease activity. Therefore, evaluation of Dickkopf-1 (Dkk-1) and secreted Frizzled related protein 5 (sFRP5), which are Wnt signaling pathway antagonists, in periodontal inflammation may be a focus of interest. A total of 99 individuals, 44 male and 55 female, participated in our study and were divided into three groups as periodontally healthy, gingivitis and periodontitis. Non-surgical periodontal treatment was applied to the disease groups. Dkk-1 and sFRP5 were evaluated in gingival crevicular fluid (GCF) at the baseline and after periodontal treatment.

DETAILED DESCRIPTION:
The participants were divided into three groups in accordance with their periodontal status according to the 2017 World Workshop on the classification of periodontal diseases : Periodontally healthy (group H, n = 33, probing depth (PD) ≤3 mm, fullmouth bleeding scores; bleeding on probing (BOP) % <10, no clinical attachment levels (CAL) and radiologic bone loss), gingivitis (group G, n = 33 PD ≤3 mm, % BOP >30, no CAL(due to periodontal disease) and radiologic bone loss), Stage 3 Grade B periodontitis (group P, n = 33, These individuals had a minimum of two non-adjacent teeth with sites with PD ≥6 mm, CAL ≥5 mm, BOP ≥30%, tooth loss due to periodontitis ≤4 teeth, the alveolar bone loss at radiographs extending to middle or apical third of the root, the presence of consistent amounts of plaque biofilm/calculus deposits commensurate with the severity of periodontal tissue breakdown, the proportion of percentage bone loss to age values were between 0.25 and 1). Panoromic and periapical radiographic examination was also performed for the diagnosis of periodontitis.

Periodontal status of each individual included in the study was determined by measuring plaque index (PI), gingival index (GI), PD, clinical attachment level (CAL) and bleeding of probing (BOP). PD and CAL were measured on six sites (mesio-buccal/ facial, mid-buccal/facial, disto-buccal/facial, mesio-lingual/palatinal, mid-lingual/palatinal, disto-lingual/palatinal) of the teeth in baseline and after periodontal treatment. Bleeding was observed up to 10 sec after the examination of probing depth and BOP score was calculated as the number of BOP-positive sites was divided the number of total sites, after multiplied with 100. Panoramic and periapical radiographs were used to determine the alveolar bone loss. All clinical measurements were recorded using a standard Williams periodontal probe.

Within 2 weeks from the screening visit, phase 1 periodontal treatment/scaling and root planing under local anesthesia using manual instruments and ultrasonic devices in a single appointment were performed and oral hygiene instructions were given to all participants with periodontitis by a single calibrated periodontist. In gingivitis and periodontally healthy groups, phase 1 periodontal treatment and oral hygiene education were given to each one. All periodontal clinical measurements recorded and gingival crevicular fluid (GCF) samples collection were at baseline and the 6-8 th week after the periodontal treatment in patients with G and P group and at one time point (baseline) in H group.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-50 years old
* Meeting the criteria for the working groups

Exclusion Criteria:

* having any systemic or metabolic diseases or insturition of effected bone metabolism,
* having bruksizm habits,
* pregnant or lactating,
* received periodontal/peri-implant treatment within the last 6 months,
* the history of antibiotics or antiinflamatuars use regularly within the last 6 months,
* having < 20 teeth (except for 3rd molars),
* smokers or consumed alcohol.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 99 patients (44 males and 55 females) between 20-50 years of age were included and were divided into three groups as follows: periodontally healthy, patients with gingivitis, and patients with stage 3 grade B periodontitis. Participants were selected from the patients who presented for periodontal treatment between March 2024 and August 2024 at Department of Periodontology, Faculty of Dentistry, Sivas Cumhuriyet University, Sivas, Turkey.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Dkk-1 and sFRP5 levels at baseline and after periodontal treatment | 6-8 weeks
  Dkk-1 and sFRP5 levels assessed by ELISA in GCF at baseline and after non-surgical periodontal treatment were the primary outcome measures.Dkk-1 and sFRP5 will be measured by ELISA technique according to the manufacturer's instructions. The sensitivity value for Dkk-1 and sFRP5 is 0.056 ng/mL and 0.059 ng/mL, respectively. Optical densities will be taken at 450 nm wavelength, and standard concentrations and corresponding optical density values and sample optical density values will be recorded. The standard curve will be drawn according to the optical densities and concentrations of standards, and the concentrations of all samples will be calculated by the linear regression equation of the obtained standard curve.Dkk-1 and sFRP5 total amount will be given in ng unit.

SECONDARY OUTCOMES:
Gingival Crevicular Fluid (GCF)Volume at baseline and after periodontal treatment | 6-8 weeks
  GCF volume will be obtained by converting the number measured on the periotron device (=periotron unit) into microliters. This value will be stated among the groups (H, G and P) and in the G and P groups after non-surgical periodontal treatment.
Gingival index (GI) at baseline and after periodontal treatment | 6-8 weeks
  The plaque index (GI) (Löe & Silness, 1963) of each individual included in the study was measured at six sites of the teeth (mesio-buccal/facial, mid-buccal/facial, disto-buccal/facial, mesio-lingual/palatinal, mid-lingual/palatinal, disto-lingual/palatinal) with a periodontal probe at baseline and after periodontal treatment (6-8 weeks) in G and P groups and recorded with a score between 0-3.
Bleeding on probing (BOP) percentage at baseline and after periodontal treatment | 6-8 weeks
  Whether there is bleeding on probing will be determined by dividing the number of positive areas by the total number of areas and multiplying by 100. It will be stated as a percentage between the groups and within the groups after non-surgical periodontal treatment (G and P).
Probing depth (PD)at baseline and after periodontal treatment | 6-8 weeks
  Pocket depth was recorded with the help of a periodontal probe at six sites of the teeth (mesio-buccal/facial, mid-buccal/facial, disto-buccal/facial, mesio-lingual/palatinal, mid-lingual/palatinal, disto-lingual/palatinal) at the beginning and after periodontal treatment, as the distance from the gingival margin to the periodontal pocket base in mm.
Plaque index (PI) at baseline and after periodontal treatment | 6-8 weeks
  The plaque index (PI) (Silness & Löe, 1964) of each individual included in the study was measured at six sites of the teeth (mesio-buccal/facial, mid-buccal/facial, disto-buccal/facial, mesio-lingual/palatinal, mid-lingual/palatinal, disto-lingual/palatinal) with a periodontal probe at baseline and after periodontal treatment (6-8 weeks) in G and P groups and recorded with a score between 0-3.
Clinical attachment levels (CAL) at baseline and after periodontal treatment | 6-8 weeks
  Clinical attachment levels were recorded at baseline and after periodontal treatment in six regions of the teeth (mesio-buccal/facial, mid-buccal/facial, disto-buccal/facial, mesio-lingual/palatinal, mid-lingual/palatinal, disto-lingual/palatinal) using a periodontal probe, from the cementoenamel junction to the base of the periodontal pocket in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Şükran Acıpınar, Principal Investigator — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be updated and shared upon completion of the study.